CLINICAL TRIAL: NCT01649739
Title: Vardenafil as add-on Therapy for Patients With Pulmonary Hypertension Treated With Inhaled Iloprost
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Mordechai Kremer, Profesor, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMCVAR1234
Record Dates: First submitted 2012-07-22; First posted 2012-07-25 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Levitra (Experimental)
  Interventions: Drug: Levitra

INTERVENTIONS:
Drug: Levitra — There is 2 dosage:10mg Twice daily and 20mg Twice daily

SUMMARY:
Patients with pulmonary arterial hypertension (PAH) suffer from breathlessness, poor quality of life and inability to function, despite medical therapy Current consensus states that combination therapy with different classes of PAH-specific therapy is likely to bring additional benefit to PAH patients. In this study we plan to study how exercise performance changes when the phosphodiesterase inhibitor vardenafil is added to patients who remain symptomatic from PAH when treated with inhaled iloprost.

Following baseline assessment, all Patients will start vardenafil 10 mg bid. If the drug is tolerated by the patients, after a two week period, up titration to 20 mg bid will be permitted, at the discretion of the investigators.

According to treatment protocol up titration will be done carefully and whenever side effects will be reported up titration will be stopped or dosage will be decreased or stopped according to the investigator judgment.

Systemic BP will be measured at baseline assessment. The patient will attend the clinic for the first dose monitoring (10 mg) and after up titration of the study drug to 20 mg.

Systemic BP will be measured at baseline assessment. The patient will attend the clinic for the first dose monitoring (10 mg) and after up titration of the study drug to 20 mg. A fall in SBP of>30 mmHg will be considered significant or any smaller value at the discretion of the investigator. BP will be measured according to the following protocol.

Pre-dose Immediately before administration of vardenafil. This will be timed approximately one hour prior to the next planned dose of iloprost.

Pre-inhalation One hour post vardenafil dose, immediately prior to iloprost inhalation.

Post-inhalation Immediately following completion of iloprost inhalation and every fifteen minutes for one hour.

Prior to discharge Two hours following the iloprost.

Later monitoring At all follow-up visits, BP will be measured.

This is an open-label study to evaluate the safety and efficacy of adding higher doses of vardenafil to inhaled iloprost over 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. All Patients must satisfy current diagnostic criteria for pulmonary artery hypertension based on their historical right heart catheter data (within 3 years of study enrollment): Mean PAP≥25mmHg at rest by a PCWP<15mmHg and by PVR >3 Wood Units.
2. Currently stable for at least 3 months with inhaled iloprost, between 5-9 doses per day, using the I-Neb device.
3. Willing and able to participate in all study follow-up procedures.
4. New York Heart Association (NYHA) Class II-IV.
5. Six minute walking distance between 100-450 meters at the baseline assessment.
6. Women of child-bearing age must demonstrate adequate contraception or undergo a pregnancy test.
7. Patients with inoperable pulmonary thromboembolic disease or congenital heart disease are eligible for inclusion.

Exclusion Criteria:

1. Functional Class NYHA Class I.
2. PAH due to left heart disease, chronic lung diseases (VC or FEV1 <60% of predicted), chronic hypoxia or chronic thromboembolic disease.
3. Acute intercurrent illness requiring hospital admission in the month proceeding screening.
4. Any non-PAH medical condition likely to interfere with participation in evaluation of study endpoints, e.g. musculoskeletal disorders.
5. Any uncontrolled or terminal non-PAH medical condition likely to interfere with completion of the study, according to the judgment of the study physician.
6. Concomitant therapy with drugs known to interact adversely with the study drug (Nitrates, alpha-adrenergic receptor antagonists, CYP3A4 inhibitors (HIV protease inhibitors, ketoconazole, itraconazole, erythromycin
7. Chronic renal failure - creatinine clearance< 50ml/min as calculated with the Cockcroft equation.
8. Current participation in another clinical trial.
9. Pregnancy or planned pregnancy during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-05 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Change in 6 minute walk or New York Heart Association functional class. | 14 weeks

SECONDARY OUTCOMES:
Changes in Pulmonary artery pressure assessed (by echo), exercise test parameters, pro-NT BNP, quality of life. Clinical worsening during study, study drop-out and adverse events during the study. | 14 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Institute,Rabin Medical Center, Petah Tikva, Israel